CLINICAL TRIAL: NCT00228176
Title: Randomized, Multicenter, Double-blind, Placebo-controlled, Two-arm Parallel Group Trial of Rimonabant 20-mg od, for Inhibition of Atherosclerosis Progression Assessed by Carotid Artery Intima-media Thickness (CIMT), in Overweight Patients With Additional Risk Factors
Brief Title: Atherosclerosis Underlying Development Assessed by Intima-Media Thickness in Patients on Rimonabant
Acronym: AUDITOR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decision taken in light of demands by certain national health authorities
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC5828; 2005-001612-49 (EudraCT Number)
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-04

CONDITIONS: Carotid Artery Plaque; Arteriosclerosis; Obesity; Metabolic Syndrome X
Keywords: Metabolic syndrome; Carotid Atherosclerosis
MeSH Terms: conditions — Carotid Stenosis; Arteriosclerosis; Obesity; Metabolic Syndrome; Carotid Artery Diseases | interventions — Rimonabant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rimonabant (Experimental): Rimonabant 20 mg once daily
  Interventions: Drug: Rimonabant
- Placebo (Placebo Comparator): Placebo (for Rimonabant) once daily.
  Interventions: Drug: Placebo (for Rimonabant)

INTERVENTIONS:
Drug: Rimonabant — Tablet, oral administration
  Other Names: SR141716; Acomplia
  Arms: Rimonabant
Drug: Placebo (for Rimonabant) — Tablet, oral administration
  Arms: Placebo

SUMMARY:
Objectives:

* Primary: To evaluate the effect of rimonabant 20-mg once daily in comparison with placebo, on the quantitative progression of atherosclerosis as assessed by carotid artery intima-media thickness (CIMT)
* Secondary: To evaluate the safety and tolerability of the above rimonabant regimen in the study population of atherosclerosis patients.

DETAILED DESCRIPTION:
This is a Phase III, prospective, multicentre, multinational, randomized, double-blind, placebo-controlled, 2-arm parallel group trial (rimonabant 20-mg od vs placebo). There will be a three-stage screening process including successively a Screening visit, a Screening CIMT and a validation of the Screening CIMT by the Imaging Core Laboratory. Patients complying with all inclusion and exclusion criteria will be randomized in one of the 2 treatment groups less than two weeks after Screening visit. Study drug (rimonabant 20 mg od or matching placebo) will be administered during 30 to 32 months. At inclusion, patients will be counseled to follow a mild hypocaloric diet, to increase their exercise level, and to stop smoking (if smokers). Glucose/lipid parameters will be assessed at Baseline and every 6 months until the Month 30 visit. CIMT will be performed at Baseline and every 6 months until final assessment at Month 30 (primary endpoint).A post-treatment follow-up visit at Month 35 will allow the collection of all adverse events and cardiovascular outcomes occurring after last study drug administration

ELIGIBILITY:
Inclusion Criteria:

* Written and signed informed consent
* Age greater than or equal to 55 years
* Abdominal obesity defined by waist circumference > 88 cm (35 inches) in women and > 102 cm (40 inches) in men
* Metabolic syndrome diagnosed on the basis of at least two of the following additional risk factors:

  1. Triglyceride level equal to or greater than 150 mg/dL
  2. HDL cholesterol less than 40 mg/dL in men or 50 mg/dL in women
  3. Fasting glucose of equal to or greater than 110 mg/dL
  4. High blood pressure defined as equal to or greater than 140 mmHg systolic and/or equal to or greater than 90 mmHg diastolic at screening visit or current treatment by antihypertensive medication.
* Ultrasonographic evidence at Screening quantitative B-mode ultrasound imaging of a minimal CIMT measurement of greater than or equal to 0.7 mm in either of the far walls of the common carotid artery, and maximal CIMT measurement less than 3 mm in any carotid artery segment.
* All 6 carotid artery segments must have ultrasound images for all CIMT measurements
* Screening CIMT recording deemed to be of acceptable CIMT image quality, and demonstrating adherence to the CIMT interrogation protocol, as determined by the Imaging Core Laboratory's assessment.

Exclusion Criteria:

* History of very low calorie diet or surgical procedures for weight loss within 6 months prior to screening visit
* Obesity of known endocrine origin
* Uncontrolled diabetes, i.e. with HbA1c > 10%
* Anticipated survival less than 27 months
* Presence of any severe medical or psychological condition, that in the opinion of the Investigator, would compromise the subject's safety or successful participation in the study
* Presence of any other condition (e.g. geographic, social, or other), actual or anticipated, that the Investigator feels would restrict or limit the subject's participation for the duration of the study
* Receipt of any investigational treatment (drug or device) within 30 days prior to Screening
* Previous participation in a rimonabant study
* Total occlusion of any carotid artery segment
* Previous history of carotid intervention
* Patient considered at high risk of carotid intervention during the next 27 months

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 661 (Actual)
Dates: Start 2005-08; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline in averaged per patient carotid artery intima-media thickness (CIMT) | Month 30

SECONDARY OUTCOMES:
First occurrence of any component of stroke/myocardial infarction (MI)/cardiovascular death | From randomization to Month 35
First occurrence of any component of stroke/MI/cardiovascular death/hospitalization for revascularization procedure, unstable angina, transient ischemic attack (TIA) | From randomization to Month 35

CONTACTS AND LOCATIONS:
Overall Officials: John JP Kastelein, MD, Study Chair — Amsterdam UMC, location VUmc
Locations (6):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Guildford Surrey, United Kingdom

REFERENCES:
- [Result] O'Leary DH, Reuwer AQ, Nissen SE, Despres JP, Deanfield JE, Brown MW, Zhou R, Zabbatino SM, Job B, Kastelein JJ, Visseren FL; AUDITOR investigators. Effect of rimonabant on carotid intima-media thickness (CIMT) progression in patients with abdominal obesity and metabolic syndrome: the AUDITOR Trial. Heart. 2011 Jul;97(14):1143-50. doi: 10.1136/hrt.2011.223446. Epub 2011 May 24. PMID 21610270